CLINICAL TRIAL: NCT03259347
Title: Eating Disorders Programs: An Indicated Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IndPrevPilot; 1R01MH086582-01A1 (NIH)
Record Dates: First submitted 2017-03-29; First posted 2017-08-23 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Body Image; Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counter-attitudinal therapy (Experimental): Counter-attitudinal therapy (CAT) is dissonance-based group intervention. CAT consists of behavioral, written, and verbal exercises in which participants discuss the costs of pursuing the thin ideal and behaviors that are used to pursue the thin ideal. The intervention is 8 sessions long (1-hr each) and is administered by a trained facilitator who uses an intervention script. Participants will be asked to complete weekly home exercises throughout the course of the intervention.
  Interventions: Behavioral: Group-based Therapy
- Educational-support group (Active Comparator): The educational support group intervention that is representative of typical treatment groups offered at universities and community settings. For the current study, the educational support group was designed to match the dissonance group on treatment modality (group-based), duration (8 1-hr sessions), and use of an intervention script administered by a trained facilitator. In the intervention sessions, participants will be provided with a basic education about eating disorders, support for themselves and fellow group members, and learn mindfulness techniques.Participants will be asked to complete weekly homework assignments.
  Interventions: Behavioral: Group-based Therapy

INTERVENTIONS:
Behavioral: Group-based Therapy — Young women with body dissatisfaction will be randomized to one of two conditions: 1) an educational-support group condition; or 2) a counter-attitudinal therapy condition. We will test if a brief dissonance-based eating disorder prevention program produces intervention effects when delivered to participants with sub-threshold and threshold eating disorders.

SUMMARY:
The purpose of this study is to assess the effectiveness of two body acceptance programs for women. Participants may experience reduction of eating pathology and prevention of future obesity and eating disorders; may derive a sense of altruism and contribution to furthering understanding of a public health problem.

ELIGIBILITY:
Inclusion Criteria:

* Participant indicates sub-threshold or threshold eating disorder.
* Participant is available to participate in the intervention sessions.
* Participants must be MRI eligible.

Exclusion Criteria:

* Participant does not indicate sub-threshold or threshold eating disorder.
* Participant is unable to attend intervention sessions.
* Participant cannot participate if MRI ineligible.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 534 (Estimated)
Dates: Start 2012-06-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Eating Disorder Diagnostic responses using the Eating Disorder Examination questionnaire at 8 weeks and 6 months | Measured at baseline, week 8, and Month 6
  Evaluate change (if any) by using the Eating Disorder Examination questionnaire at the 8 week and 6 month mark.

SECONDARY OUTCOMES:
Assessments using Ideal-Body Stereotype Scale-Revised | Measured at baseline, week 8, and Month 6
  Evaluate the participants' perception of the ideal-body stereotype
Assessments using Satisfaction and Dissatisfaction with Body Parts Scale | Measured at baseline, week 8, and Month 6
  Evaluate participants' level of satisfaction and dissatisfaction with specific parts of their bodies
Assessments using Dutch Restrained Eating Scale | Measured at baseline, week 8, and Month 6
  Evaluate participants ability to exercise restraint in regards to food
Assessments using Positive Affect and Negative Affect Scale-Revised | Measured at baseline, week 8, and Month 6
  Measure participants' affect and monitor any changes that may occur.
Assessments using Beliefs About Appearance Scale | Measured at baseline, week 8, and Month 6
  Evaluate participants' perceptions and beliefs on physical appearance.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Oregon Research Institute, Eugene, Oregon
  - Drexel University, Philadelphia, Pennsylvania
  - The University of Texas, Austin, Texas

REFERENCES:
- [Derived] Stice E, Rohde P, Shaw H, Gau JM. Randomized trial of a dissonance-based group treatment for eating disorders versus a supportive mindfulness group treatment. J Consult Clin Psychol. 2019 Jan;87(1):79-90. doi: 10.1037/ccp0000365. PMID 30570303